CLINICAL TRIAL: NCT02432859
Title: The Effect of Electrical Stimulation on the Expression of VEGF, VEGFR-2, HIF and NO in the Diabetic Foot Ulcer
Brief Title: Electrical Stimulation and Expression of VEGF, VEGFR-2, HIF and NO in the Diabetic Foot Ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarbiat Modarres University (Other)
Responsible Party: Principal Investigator, giti torkaman, Professor of physical therapy, Physical therapy department, Faculty of medical sciences, Tarbiat modares univercity, Tarbiat Modarres University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D52/2509
Record Dates: First submitted 2015-04-16; First posted 2015-05-04 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot | interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electrical stimulation (Active Comparator): In the electrical stimulation group, group who received direct current ES at sensory threshold intensity for 1 h/day, 3 days/week, for 4 weeks (12 sessions)
  Interventions: Procedure: Electrical Stimulation
- Placebo (Placebo Comparator): In the placebo group, the treatment procedure was the same as that the ES group, but the current intensity was zero
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Electrical Stimulation — Direct current with sensory intensity for one hour
  Other Names: Direct current ES
  Arms: Electrical stimulation
Procedure: Placebo — Direct current with zero intensity for one hour
  Other Names: Placebo Direct current ES
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether electrical stimulation is effective in the expression of VEGF, VEGFR-2, HIF-1α and NO and healing in diabetic foot ulcer.

DETAILED DESCRIPTION:
30 type 2 diabetic patients with ischemic foot ulceration were enrolled. Patients were randomly assigned to electrical stimulation (ES, n=15) or sham ES (placebo, n=15) groups. ES group received cathodal direct current for 1 h/day, 3 days/week, for 4 weeks (12 sessions). Wound fluid sample was collected for VEGF, VEGFR-2, HIF-1α and NO measurement in the first and last treatment sessions before and after intervention. Wound surface area (WSA) was measured at 1st, 6th, and 12th session.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic diabetic foot ulcer
* Wagner classification DFU 2
* 0.5<ABI<0.9
* Mild to moderate diabetic neuropathy

Exclusion Criteria:

* Fracture in a lower limb
* A severe infection
* A malignancy
* Kidney failure
* Skin diseases
* Osteomyelitis
* Pregnancy

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-11; Primary Completion 2014-09 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
The wound fluid level of VEGF, VEGFR-2, HIF-1α and NO (pg/ml) | Change from Baseline in wound fluid level of VEGF, VEGFR-2, HIF-1α and NO at 4 weeks

SECONDARY OUTCOMES:
Wound surface area(cm2) | Change from Baseline in wound surface area at 2 and 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Giti Torkaman, PhD, Study Director — Professor of Physical Therapy, Physical Therapy Department, Faculty of Medical Sciences, Tarbiat Modares Univercity
Locations (1):
- Tarbiat Modares University, Tehran, Iran